CLINICAL TRIAL: NCT00599976
Title: Randomized Controlled Trial of Pulmonary Vein Antrum Isolation vs. AV Node Ablation With Bi-Ventricular Pacing for Treatment of Atrial Fibrillation in Patients With Congestive Heart Failure (PABA CHF)
Brief Title: Comparison of Pulmonary Vein Isolation Versus AV Nodal Ablation With Biventricular Pacing for Patients With Atrial Fibrillation With Congestive Heart Failure (PABA CHF)
Acronym: PABA CHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Policlinico Umberto I (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Andrea Natale, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA 007; No 757, ME 836 Czech Republic.
Record Dates: First submitted 2008-01-02; First posted 2008-01-24 (Estimated); Last update posted 2008-01-24 (Estimated); Status verified 2007-12

CONDITIONS: Atrial Fibrillation; Congestive Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Pulmonary vein isolation — Pulmonary vein isolation
  Other Names: atrial fibrillation ablation

SUMMARY:
For patients with atrial fibrillation and heart failure, current treatment can include AV nodal ablation with biventricular pacing. Pulmonary vein isolation (PVI) is a new procedure for this patient population which attempts to restore sinus rhythm. This trial is a randomized controlled trial of AVN ablation with biventricular pacing versus PVI for atrial fibrillation patients with congestive heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic atrial fibrillation with NYHA II-III symptoms despite the use of anti-arrhythmic medications.
* Ejection fraction was required to be ≤ 40%.
* Patients were required to be on a heart failure regimen that included beta-blockers and ace-inhibitors or angiotensin receptor blockers for all patients and spironolactone for NYHA III patients.
* Patients were required to complete a 6-minute walk test and to be ≥ 18 years of age.

Exclusion Criteria:

* Reversible causes of AF and heart failure (HF) such as pericarditis, hyperthyroidism, valvular heart disease and tachycardia-induced cardiomyopathy.
* Post-operative AF, previous MAZE or MAZE-like surgery, previous left atrial instrumentation
* Life expectancy ≤ 2 years
* Likely cardiac transplant within the next 12 months
* Contraindication to anti-arrhythmic medications and/or anticoagulation
* Severe pulmonary disease
* Documented intra-atrial thrombus
* Tumor or other abnormalities which preclude catheter introduction
* Cardiac surgery, MI or PCI within the past three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2002-11; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
composite of EF, 6-minute walk distance and MLWHF score | 6 months

SECONDARY OUTCOMES:
freedom from AF and left atrial size | 6 months

REFERENCES:
- [Derived] Khan MN, Jais P, Cummings J, Di Biase L, Sanders P, Martin DO, Kautzner J, Hao S, Themistoclakis S, Fanelli R, Potenza D, Massaro R, Wazni O, Schweikert R, Saliba W, Wang P, Al-Ahmad A, Beheiry S, Santarelli P, Starling RC, Dello Russo A, Pelargonio G, Brachmann J, Schibgilla V, Bonso A, Casella M, Raviele A, Haissaguerre M, Natale A; PABA-CHF Investigators. Pulmonary-vein isolation for atrial fibrillation in patients with heart failure. N Engl J Med. 2008 Oct 23;359(17):1778-85. doi: 10.1056/NEJMoa0708234. PMID 18946063